CLINICAL TRIAL: NCT06297434
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase IIa Clinical Trial to Evaluate the Safety and Explore the Efficacy of J2H-1702 for Non-alcoholic Steatohepatitis
Brief Title: Phase 2a Study to Evaluate Safety and Explore Efficacy of J2H-1702 for NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: J2H Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JH-221-201
Record Dates: First submitted 2024-02-13; First posted 2024-03-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- J2H-1702 A mg (Experimental)
  Interventions: Drug: J2H-1702
- J2H-1702 B mg (Experimental)
  Interventions: Drug: J2H-1702
- J2H-1702 C mg (Experimental)
  Interventions: Drug: J2H-1702
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: J2H-1702 — Orally, once daily before meals
  Arms: J2H-1702 A mg
Drug: J2H-1702 — Orally, once daily before meals
  Arms: J2H-1702 B mg
Drug: J2H-1702 — Orally, once daily before meals
  Arms: J2H-1702 C mg
Drug: Placebo — Orally, once daily before meals
  Arms: Placebo

SUMMARY:
The study aims to evaluate the safety of J2H-1702 compared to the placebo and explore the efficacy of J2H-1702 at Week 12 timepoint after administration compared to baseline in patients with NASH.

DETAILED DESCRIPTION:
Subjects will be randomized to the study group 1 (J2H-1702 A mg), study group 2 (J2H-1702 B mg), study group 3 (J2H-1702 C mg), or control group (placebo of J2H-1702) in a 1:1:1:1 ratio and administered the investigational product (IP) for 12 weeks. After the IP administration, the safety and efficacy will be evaluated at V4, V8 and V12 (end of treatment, EOT).

ELIGIBILITY:
Inclusion Criteria:

1. A subject aged ≥19 years to ≤75 years
2. Meeting all of the following criteria:

   * Screening MRI-PDFF with ≥8% steatosis
   * Screening MRE with liver stiffness ≥2.5 kPa
   * ALT or AST ≤250 IU/L at screening
3. Willing to maintain the same lifestyle (exercise, alcohol consumption, diet, etc.) during the study
4. Voluntarily provide written consent to participate in the study

Exclusion Criteria:

1. A subject who has past or current history of liver diseases
2. A subject who has the following medical or surgical history

   * Severe cardiac diseases, Malignant tumors, Clinically significant hypersensitivity reaction to any drugs containing components of the 11β-HSD1 inhibitor or same class
3. A subject who has the following concomitant diseases

   * liver disease, uncontrolled hypertension, uncontrolled DM, etc.
4. A subject who has taken the following medications

   * Systemic glucocorticoids, NSAIDs, any medication that may induce fatty liver disease, etc.
5. A subject who has taken IP of another study
6. A subject who does not agree with appropriate methods of contraception

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in results on MRI-PDFF at week12. | Baseline and week12
  The liver fat content(%) on MRI-PDFF at week 12 after administration of the IP are evaluated.
Changes from baseline in results on MRE at week12. | Baseline and week12
  The liver fibrosis (kPa) on MRE at week 12 after administration of the IP are evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- J2H Biotech, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No